CLINICAL TRIAL: NCT01967732
Title: A Single-center, Open-label, Randomized, Controlled, Crossover Study to Investigate the Nicotine Pharmacokinetic Profile and Safety of Tobacco Heating System 2.2 (THS 2.2) Following Single Use in Smoking, Healthy Subjects Compared to Conventional Cigarettes and Nicotine Nasal Spray.
Brief Title: Nicotine Pharmacokinetic Profile and Safety of the Tobacco Heating System 2.2 (THS 2.2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZRHR-PK-01-EU; ZRHR-PK-01-EU (Other: Philip Morris Products S.A.); 2013-003097-27 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Smoking; Nicotine absorption; Modified risk tobacco product; Conventional cigarette; Nicotine replacement therapy; Nicotine nasal spray
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- THS 2.2 then CC (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of THS 2.2)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of CC).
  Interventions: Other: THS 2.2; Other: CC
- CC then THS 2.2 (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of CC)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of THS 2.2).
  Interventions: Other: THS 2.2; Other: CC
- THS 2.2 then NNS (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of THS 2.2)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single administration of NNS)
  Interventions: Other: THS 2.2; Other: NNS
- NNS then THS 2.2 (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single administration of NNS)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of THS 2.2).
  Interventions: Other: THS 2.2; Other: NNS

INTERVENTIONS:
Other: THS 2.2 — Single use of the Tobacco Heating System 2.2 (THS 2.2)
Other: CC — Single use of subject's own conventional cigarette (CC)
  Arms: CC then THS 2.2; THS 2.2 then CC
Other: NNS — Single administration of 1 mg of nicotine
  Arms: NNS then THS 2.2; THS 2.2 then NNS

SUMMARY:
The primary objective of this clinical study is to evaluate the pharmacokinetic (PK) profile (rate and amount of nicotine absorbed) following a single use of the THS 2.2 compared to the PK profiles from a single use of a conventional cigarette (CC) and from a single use of nicotine nasal spray (NNS).

ELIGIBILITY:
Inclusion Criteria:

* Subject is Caucasian
* Smoking, healthy subject as judged by the Investigator.
* Subject has smoked at least 10 commercially available non menthol CCs per day (no brand restrictions) for the last 4 weeks.
* Subject has smoked for at least the last 3 consecutive years.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of a drug (whichever is longer) which has an impact on CYP2A6 activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Adrian Johnston Stewart, MD, Principal Investigator — Celerion GB Ltd.
Locations (1):
- Celerion GB Ltd, 22-24 Lisburn Road, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 01 November 2013
  At admission (Day -1), all the subjects performed a product trial (THS 2.2 and subsequently NNS).
  From enrollment, they were asked to remain abstinent from smoking for at least 24 hours (Day 0) before being randomized on Day 1 into 1 of the 4 sequences.
Pre-assignment Details: Enrolled population = 62 subjects = 62 randomized as described below:
  * Sequence "THS 2.2 then CC": 22 subjects
  * Sequence "CC then THS 2.2": 22 subjects
  * Sequence "THS 2.2 then NNS": 9 subjects
  * Sequence "NNS then THS 2.2": 9 subjects
Period: Washout Period of 1 Day (Day 0)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NNS | NNS Then THS 2.2
Started | 22 | 22 | 9 | 9
Completed | 22 | 21 | 9 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Dropped due to personal reasons | 0 | 1 | 0 | 0
Period: First Intervention (Day 1)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NNS | NNS Then THS 2.2
Started | 22 | 21 | 9 | 9
Completed | 22 | 20 (Subject discontinued from the study prior to product use) | 9 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Poor venous access | 0 | 1 | 0 | 0
Period: Washout Period of 1 Day (Day 2)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NNS | NNS Then THS 2.2
Started | 22 | 20 | 9 | 9
Completed | 22 | 20 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (Day 3)
Arm/Group | THS 2.2 Then CC | CC Then THS 2.2 | THS 2.2 Then NNS | NNS Then THS 2.2
Started | 22 | 20 | 9 | 9
Completed | 22 | 20 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: PK population: all randomized subjects who completed at least 1 of the single-use days, with at least 1 derived PK parameter. No subjects were excluded due to major protocol deviations impacting the evaluation of the results.
  62 randomized: 44 in Group 1, 18 in Group 2
  60 completers: 42 in Group 1 (2 discontinued), 18 in Group 2
Groups:
- Group 1: This population comprises the following sequences:
  * Sequence "THS 2.2 then CC"
  * Sequence "CC then THS 2.2"
- Group 2: This population comprises the following sequences:
  * Sequence "THS 2.2 then NNS"
  * Sequence "NNS then THS 2.2"
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 42 | 18 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.98) | 30.6 (5.80) | 31.7 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 25 | 10 | 35
International Organization for Standardization (ISO) nicotine level [Number; unit: participants]
  ≤ 0.6 mg | 17 | 8 | 25
  > 0.6 to ≤ 1 mg | 25 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of THS 2.2, CC and NNS
Description: Derived from multiple blood sampling on Day 1 and Day 3 (1 blood sampling pre-product use and multiple blood sampling over 24 hours post-product use).
  Geometric Least Squares means are provided.
Time Frame: 3 days
Population: PK populations consisted of all the randomized subjects who completed at least 1 of the single use days (Days 1 or 3), and for whom at least 1 PK parameter could be derived. Subjects with major protocol deviations that impacted the evaluability of the results were excluded from the PK populations.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- THS 2.2 - Group 1; CC - Group 1: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "THS 2.2 then CC"
  * Sequence "CC then THS 2.2"
- THS 2.2 - Group 2; NNS - Group 2: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "THS 2.2 then NNS"
  * Sequence "NNS then THS 2.2"
Arm/Group | THS 2.2 - Group 1 | CC - Group 1 | THS 2.2 - Group 2 | NNS - Group 2
Number analyzed (Participants) | 42 | 42 | 18 | 18
ng/mL | 9.62 [8.28 to 11.17] | 12.42 [10.69 to 14.42] | 10.52 [7.91 to 13.98] | 3.51 [2.63 to 4.66]
Statistical Analysis 1: Comparison: THS 2.2 - Group 1 vs CC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of THS 2.2:CC) for Cmax, therefore, there was no statistical hypothesis to be tested for this objective; Test type: Superiority or Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 77.43, 95% CI 2-sided [62.69 to 95.63] — LS mean ratio (THS 2.2 - Group 1:CC - Group 1)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (Pre-product Use) to Last Time Point [AUC(0-last)] Following Single Use of THS 2.2, CC and NNS
Description: as for outcome 1
Time Frame: 3 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | THS 2.2 - Group 1 | CC - Group 1 | THS 2.2 - Group 2 | NNS - Group 2
Number analyzed (Participants) | 42 | 42 | 18 | 18
h*ng/mL | 15.10 [13.19 to 17.29] | 20.28 [17.71 to 23.22] | 17.87 [13.79 to 23.15] | 8.02 [6.19 to 10.39]
Statistical Analysis 1: Comparison: THS 2.2 - Group 1 vs CC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of THS 2.2:CC) for AUC(0-last), therefore, there was no statistical hypothesis to be tested for this objective; Test type: Superiority or Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 74.47, 95% CI 2-sided [61.52 to 90.14] — LS mean ratio (THS 2.2 - Group 1:CC - Group 1)

ADVERSE EVENTS:
Time Frame: From the informed consent form (ICF( signature until the end of the safety follow-up period (7 days after discharge of the subject)
Description: The safety was assessed in the safety population, consisting of 62 subjects: 44 subjects in Group 1, 18 subjects in Group 2. This population includes all the subjects exposed to THS 2.2 and NNS from the product trials on Day -1.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/18
Other Adverse Events (participants affected / at risk) | 15/44 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=44) | Group 2 (N=18)
Dizziness (Nervous system disorders) | 6 (7) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Presyncope (Nervous system disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2014-08-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT01967732/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT01967732/SAP_001.pdf